CLINICAL TRIAL: NCT06707610
Title: A First-in-Human, Open-Label, Multi-Center Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antitumor Activity of ALK202 for Injection in Adult Participants with Advanced Solid Tumors
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics (PK), and Antitumor Activity of ALK202 in Participants with Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Allink Biotherapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ALK202-01
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Advanced Cancer; Advanced Solid Tumor
Keywords: First-in-human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Part A: Dose-escalation Phase Part B: Dose-expansion Phase (Experimental): A dose-escalation study to determine the MTD and the subsequent doses for dose expansion study (Part B). A dose-expansion study which will enroll the select indications.
  Interventions: Drug: ALK202

INTERVENTIONS:
Drug: ALK202 — Administered intravenously, once every 3 weeks

SUMMARY:
TThis is a first-in-human (FIH), open-label, multicenter dose escalation and expansion study of ALK202. The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (PK), and antitumor activity of ALK202 as a monotherapy in adult participants with Advanced Solid Tumors. The study will also identify recommended dose(s) for subsequent clinical studies of ALK202.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥18 and ≤75 years old on the day of signing the ICF
* At least 1 measurable lesion per RECIST v1.1
* Expected survival ≥3 months
* ECOG PS score of 0 or 1
* Adequate organ function
* Female participants of childbearing potential or male participants whose partner is a female of childbearing potential agree to use medically effective contraceptive methods (abstinence, birth control pills, barrier contraception, intra-uterine contraceptive device, etc.) from the date of signing the ICF until at least 6 months after the last dose of ALK202, and during this period, male participants are not allowed to donate sperms.

Exclusion Criteria:

* Received organ transplant or hematopoietic stem cell transplant previously
* Vaccinated with live vaccines within 4 weeks prior to the first dose
* Primary central nervous system malignancies, or active metastases to central nervous system and/or metastases to meninges
* Pregnant or lactating women
* Pleural effusion, pericardial effusion, or intraperitoneal effusion accompanied with clinical symptoms, clinically poorly controlled, or requiring repeated drainage.
* Evidence of other severe or uncontrolled systemic diseases (e.g., decompensated respiratory disorder, hepatic disease, or renal disease).

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of ALK202 in adult participants with advanced solid tumors; To determine the maximum tolerated dose (MTD); To determine the recommended dose(s) of ALK202 for subsequent clinical studies. | Approximately 36 months
  Dose-limiting toxicity (DLT); The incidence and severity of treatment-emergent adverse events (TEAEs) and treatment-related adverse events (TRAEs) according to CTCAE v5.0.

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics (PK) of ALK202 | Approximately 36 months
  PK parameters after single and multiple doses: area under the concentration-time curve from time zero to the last measurement (AUC0-last)
To evaluate the pharmacokinetics (PK) of ALK202 | Approximately 36 months
  PK parameters after single and multiple doses: area under the concentration-time curve from time zero to infinity (AUC0-inf)
To evaluate the pharmacokinetics (PK) of ALK202 | Approximately 36 months
  PK parameters after single and multiple doses: Maximum serum Concentration (Cmax)
To evaluate the pharmacokinetics (PK) of ALK202 | Approximately 36 months
  PK parameters after single and multiple doses: Time to Maximum Concentration(Tmax)
To evaluate the pharmacokinetics (PK) of ALK202 | Approximately 36 months
  PK parameters after single and multiple doses: trough Concentration(Ctrough)
To evaluate the pharmacokinetics (PK) of ALK202 | Approximately 36 months
  PK parameters after single and multiple doses: Clearance(CL)
To evaluate the pharmacokinetics (PK) of ALK202 | Approximately 36 months
  PK parameters after single and multiple doses: apparent Distribution Volume(Vd)
To evaluate the pharmacokinetics (PK) of ALK202 | Approximately 36 months
  PK parameters after single and multiple doses: steady-state apparent distribution volume (Vss)
To evaluate the pharmacokinetics (PK) of ALK202 | Approximately 36 months
  PK parameters after single and multiple doses: terminal half-life (t1/2)
To evaluate the immunogenicity of ALK202 | Approximately 36 months
  The generation of anti-drug antibodies (ADAs)
To evaluate the preliminary antitumor activity of ALK202 | Approximately 36 months
  Objective Response Rate (ORR)
To evaluate the preliminary antitumor activity of ALK202 | Approximately 36 months
  Duration of Response (DOR)
To evaluate the preliminary antitumor activity of ALK202 | Approximately 36 months
  Disease Control Rate (DCR)
To evaluate the preliminary antitumor activity of ALK202 | Approximately 36 months
  Progression-Free Survival (PFS)
To evaluate the preliminary antitumor activity of ALK202 | Approximately 36 months
  Overall Survival (OS)
To evaluate the biomarkers | Approximately 36 months
  To explore the correlation between biomarkers (EGFR/c-MET) and the efficacy and other clinical outcomes/parameters of ALK202

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - D&H Cancer Research Center Llc, Margate, Florida
  - Next Oncology, Fairfax, Virginia
- Australia (2):
  - Scientia Clinical Research Ltd, Randwick, New South Wales
  - Macquarie University, Sydney, New South Wales

IPD SHARING:
Plan to Share IPD: Undecided